CLINICAL TRIAL: NCT06322667
Title: A Multicenter, Postmarketing Observational Study to Evaluate Safety Regarding Amyloid-Related Imaging Abnormalities and Their Management in Patients With Early Alzheimer's Disease and Treated With Lecanemab
Brief Title: A Post Marketing Study in Participants With Early Alzheimer's Disease Treated With Lecanemab
Status: Recruiting | Type: Observational
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Other Study IDs: BAN2401-J081-401
Record Dates: First submitted 2024-03-14; First posted 2024-03-21 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Alzheimer's Disease
Keywords: Early Alzheimer's Disease; Lecanemab; ARIA
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All Participants: Participants prescribed lecanemab by a physician in routine clinical practice (post-marketing surveillance) will be observed prospectively for up to a maximum of 156 weeks or to the time of discontinuation, whichever occurs first.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — This is a non-interventional study.

SUMMARY:
The primary purpose of this study is to investigate the characteristics of amyloid related imaging abnormalities (ARIA) and investigate the treatment continuation status (e.g., continuation, interruption) after the onset of ARIA in routine clinical practice in participants treated with lecanemab.

ELIGIBILITY:
Inclusion Criteria:

* All participants who are treated with lecanemab in routine clinical practice

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants prescribed lecanemab by a physician in routine clinical practice.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2024-02-14 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Amyloid Related Imaging Abnormality-Oedema/Effusion (ARIA-E) and Amyloid Related Imaging Abnormality-Microhemorrhage and Hemosiderin Deposit, and Cerebellar Microhaemorrhage (ARIA-H) | Up to 156 weeks
Number of Participants With Interruption or Discontinuation of Lecanemab After Onset of ARIA | Up to 156 weeks

SECONDARY OUTCOMES:
Number of Participants With Infusion Related Reaction | Up to 156 weeks

CONTACTS AND LOCATIONS:
Locations (3):
- Japan (3):
  - Eisai trial site 2, Hiroshima
  - Eisai trial site 3, Kyoto
  - Eisai trial site 1, Tokyo

IPD SHARING:
Plan to Share IPD: Yes
Eisai's data sharing commitment and further information on how to request data can be found on our website http://eisaiclinicaltrials.com/.